CLINICAL TRIAL: NCT00567242
Title: Treating Intention In Aphasia: Neuroplastic Substrates
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DC007387-01A1 (NIH); R01DC007387 (NIH)
Record Dates: First submitted 2007-11-30; First posted 2007-12-04 (Estimated); Results first posted 2012-05-01 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-04

CONDITIONS: Aphasia; Cerebrovascular Accident
Keywords: aphasia; therapies, investigational; rehabilitation of speech and language disorders; magnetic resonance imaging, functional; language
MeSH Terms: conditions — Aphasia; Stroke; Language Disorders; Language

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Word-finding with intention component (Experimental): Treats word-finding (picture naming, category member generation) with an intention manipulation (complex left-hand movement to initiate word-finding trials)
  Interventions: Behavioral: Word-finding with intention component
- Word-finding with no intention component (Active Comparator): Word-finding trials similar to intention mediated treatment, but without intention manipulation
  Interventions: Behavioral: Word-finding with no intention component

INTERVENTIONS:
Behavioral: Word-finding with intention component — Word-finding trials (picture-naming) with intention manipulation (initiating word-finding trials with a complex left-hand movement). 8 (or more) baseline sessions over 4 days followed by 30 treatment sessions (2 sessions/day, 5 days/week for 3 weeks).
  Other Names: Intention Treatment
  Arms: Word-finding with intention component
Behavioral: Word-finding with no intention component — Word-finding trials with no intention manipulation. 8 (or more) baseline sessions in 4 days followed by 30 treatment sessions (2 sessions/day, 5 days/week for 3 weeks).
  Other Names: Control Treatment
  Arms: Word-finding with no intention component

SUMMARY:
The purpose of this study is to determine if an "intentional act" improves treatment response for patients with nonfluent aphasia. The treatment involves naming pictures and saying members of categories. The "intentional act" requires initiating picture naming or category member trials with a left-hand movement sequence. Nonfluent aphasia is a disorder of language production in which patients with damage to the brain's language system have trouble initiating and maintaining spoken communication. All patients participating in the study take part in functional MRI scans to determine how treatments affect brain systems.

DETAILED DESCRIPTION:
A new treatment manipulating intention substrates for language production in "nonfluent" aphasia patients was developed. The intention component involves initiating word-finding trials with a complex left-hand movement. The study addresses (1) whether or not the intention manipulation (complex left-hand movement) makes a unique contribution to treatment outcome and (2) whether or not the intention manipulation helps to shift word production mechanisms from the left to the right frontal lobe. All study participants take part in functional magnetic resonance imaging (fMRI) scans of word-finding before and after treatment and at 3-month follow-up to measure changes in lateralization of frontal lobe activity during word finding. Only patients with a substantial degree of left frontal activity on the pre-treatment fMRI scan can participate. There are three specific aims: (1) to determine if repetitive initiation of word production with a complex left-hand movement leads to increased right-hemisphere lateralization of frontal activity and if these changes can be attributed to the intention component of treatment, (2) to determine whether activity in posterior perisylvian cortices that is entrained to right frontal activity shows a greater increase in right-hemisphere lateralization from pre- to post-treatment fMRI when the intention component is included in treatment, and (3) to determine whether onset of hemodynamic responses (HDRs) in right motor/premotor cortex becomes more closely associated with the temporal onset of participants' spoken responses across treatment when the intention component is included in treatment. If successful, the treatment can provide a new treatment vehicle for increasing language function in patients with "nonfluent" aphasia.

ELIGIBILITY:
Inclusion Criteria:

* Nonfluent aphasia caused by stroke
* Moderate to severe word-finding problems
* 6 or more months post stroke
* Right handed prior to stroke
* All strokes in left hemisphere
* Native English speaker
* Capable of following verbal directions

Exclusion Criteria:

* Severe impairment of word comprehension
* Brain injury or disease in addition to stroke
* Drug or alcohol abuse within past 6 months
* Schizophrenia or other psychiatric disorder necessitating hospitalization
* History of learning disability
* Claustrophobia
* Cardiac pace-maker
* Ferrous metal implants not attached to bone, metal fragments in body
* Profound hearing loss

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Crosson, PhD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - University of Florida/Shands Hospital, Jacksonville, Florida
  - Brooks Center for Rehabilitation Studies, Jacksonville, Florida

REFERENCES:
- [Background] Crosson B, Fabrizio KS, Singletary F, Cato MA, Wierenga CE, Parkinson RB, Sherod ME, Moore AB, Ciampitti M, Holiway B, Leon S, Rodriguez A, Kendall DL, Levy IF, Rothi LJ. Treatment of naming in nonfluent aphasia through manipulation of intention and attention: a phase 1 comparison of two novel treatments. J Int Neuropsychol Soc. 2007 Jul;13(4):582-94. doi: 10.1017/S1355617707070737. Epub 2007 May 18. PMID 17521480
- [Background] Crosson B, McGregor K, Gopinath KS, Conway TW, Benjamin M, Chang YL, Moore AB, Raymer AM, Briggs RW, Sherod MG, Wierenga CE, White KD. Functional MRI of language in aphasia: a review of the literature and the methodological challenges. Neuropsychol Rev. 2007 Jun;17(2):157-77. doi: 10.1007/s11065-007-9024-z. Epub 2007 May 25. PMID 17525865
- [Background] Gopinath K, Crosson B, McGregor K, Peck K, Chang YL, Moore A, Sherod M, Cavanagh C, Wabnitz A, Wierenga C, White K, Cheshkov S, Krishnamurthy V, Briggs RW. Selective detrending method for reducing task-correlated motion artifact during speech in event-related FMRI. Hum Brain Mapp. 2009 Apr;30(4):1105-19. doi: 10.1002/hbm.20572. PMID 18465746
- [Background] Conway T, Heilman KM, Gopinath K, Peck K, Bauer R, Briggs RW, Torgesen JK, Crosson B. Neural substrates related to auditory working memory comparisons in dyslexia: an fMRI study. J Int Neuropsychol Soc. 2008 Jul;14(4):629-39. doi: 10.1017/S1355617708080867. PMID 18577292

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from December 2006 through August 2009. Fourteen subjects with minimally nonfluent aphasia, anomia, and at least some degree of frontal lesion participated in the study.
Pre-assignment Details: Prior to trial assignment, subjects underwent a functional MRI scan to determine degree of lateralization of frontal activity during word generation. Subjects with a high degree of right frontal lateralization of activity were excluded. Further, patients whose naming scores indicated that they were no more than minimally anomic were excluded.
Groups:
- Word-finding With Intention Manipulation: Treats word-finding (picture naming, category member generation) with an intention manipulation (complex left-hand movement to initiate word-finding trials)
- Word-finding With no Intention Manipulation: Word-finding trials similar to intention mediated treatment, but without intention manipulation
Period: Overall Study
Arm/Group | Word-finding With Intention Manipulation | Word-finding With no Intention Manipulation
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Word-finding With Intention Manipulation | Word-finding With no Intention Manipulation | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 7
  >=65 years | 5 | 2 | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 70.86 (12.35) | 63.00 (9.22) | 66.93 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Lateralization of Frontal Lobe (and Posterior Perisylvian) Activity During Word Production
Description: Functional MRI laterality indices (LIs)were calculated for lateral frontal, medial frontal, and posterior perisylvian cortex regions of interest (ROIs): L=number of active voxels in left hemisphere ROI and R=number of active voxels in right hemisphere ROI using the following formula: (L-R)/(L+R). LIs could vary from -1 (completely right lateralized) to +1 (completely left lateralized). Then, change in LIs was calculated by subtracting the pre-treatment from the post-treatment and 3-mo follow-up LI. It was expected the intention manipulation would show a rightward shift in LI.
Time Frame: immediately post-treatment scan minus pre-treatment baseline scan
Population: Data for all subjects completing the protocol for their respective arm were analyzed.
Measure: Mean (Standard Deviation); unit: laterality index
Arm/Group | Word-finding With Intention Manipulation | Word-finding With no Intention Manipulation
Number analyzed (Participants) | 7 | 7
laterality index | -0.2802 (0.1077) | -0.1832 (0.2768)
Statistical Analysis 1: Comparison: Word-finding With Intention Manipulation; H1: The Intention Group will show a significant rightward shift in lateral frontal laterality from pre-treatment to post-treatment. H0: The Intention Group will show no shift in lateral frontal laterality from pre-treatment to post-treatment. Since this is a repeated measures t test, the data are presented as the mean and standard deviation for for the post-treatment laterality index minus the pre-treatment laterality index; Test type: Superiority or Other; p < .05, t-test, 1 sided; Mean Difference (Final Values) = -0.2801, 95% CI 1-sided [upper limit -0.0709], Standard Error of Mean 0.1077
Statistical Analysis 2: Comparison: Word-finding With no Intention Manipulation; H1: The Control Group will show a significant rightward shift in lateral frontal lateral indices from pre-treatment to post-treatment. H0: The Control group will show no shift in lateral frontal laterality indices from pre-treatment to post-treatment. Since the analysis to test these hypotheses is a repeated-measures t-test, the mean and standard deviation are given for post-treatment laterality index minus pre-treatment laterality index; Test type: Superiority or Other; p < .05, t-test, 1 sided; Mean Difference (Final Values) = -0.1832, 95% CI 1-sided [upper limit 0.3546], Standard Error of Mean 0.2768

2. Secondary Outcome: Picture Naming Probe Scores (% Accuracy)
Description: Improvement for the time series from 8 baseline sessions through 30 treatment sessions for naming probes was computed with the C statistic using Tryon's (1982, 1983) formula for each subject. C statistics were converted to Z scores, using the formula provided by Tryon (1982). Z scores indicated treatment change for each subject, with a positive and significant Z score indicating substantive treatment gains. Z scores were then compared between groups with a t statistic. It was expected that the intention manipulation would lead to greater treatment gains than when it was not used.
Time Frame: trend for time series of 8 baseline + 30 treatment sessions
Population: Data from all subjects completing their respective arms were analyzed, with the exception that one control subject was eliminated because of an unstable baseline measure.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Word-finding With Intention Manipulation | Word-finding With no Intention Manipulation
Number analyzed (Participants) | 7 | 6
Z score | 3.68 (1.61) | 3.92 (1.18)
Statistical Analysis 1: Comparison: Word-finding With Intention Manipulation vs Word-finding With no Intention Manipulation; H1: The Intention Group would show more improvement across treatment than the Control Group. H0: The Intention Group and the Control Group would not show any difference in improvement across treatment; Test type: Superiority or Other; p < .05, t-test, 1 sided; Median Difference (Final Values) = -0.24, 95% CI 1-sided [lower limit -1.81], Standard Error of Mean 0.88

3. Secondary Outcome: Category Member Generation Probe Scores (% Accuracy)
Description: as for outcome 2
Time Frame: trend for time series of 8 baseline + 30 treatment sessions
Population: Data from all subjects completing their respective arms were analyzed, with the exception of one control subject whose baseline was not stable.
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Word-finding With Intention Manipulation | Word-finding With no Intention Manipulation
Number analyzed (Participants) | 7 | 6
Z score | 3.50 (0.83) | 1.94 (1.75)
Statistical Analysis 1: Comparison: Word-finding With Intention Manipulation vs Word-finding With no Intention Manipulation; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < .05, t-test, 1 sided; Mean Difference (Final Values) = 1.56, 95% CI 1-sided [lower limit 0.26], Standard Error of Mean 0.73

ADVERSE EVENTS:
Time Frame: Baseline to 3-month follow-up
Arm/Group | Word-finding With Intention Manipulation | Word-finding With no Intention Manipulation
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

LIMITATIONS AND CAVEATS:
1. Patients who had aphasia were enrolled. Groups were equated for anomia severity, but not type of aphasia. Aphasia types were not evenly distributed between groups which may affect results.
2. Intention subjects were older than Control Subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No